CLINICAL TRIAL: NCT07034833
Title: Assessment of a Ventriloquist Puppet for Reducing Dental Anxiety in Children
Acronym: Puppets
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hamdy Badreldin, lecturer of pediatric dentistry and oral health, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1200/384
Record Dates: First submitted 2025-05-22; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; behavior management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group: 25 child managed by basic behavior management tecniques (No Intervention): this group managed normaly with the basic behavior managment techniques like tell , show , do and others
- puppet therapy group: Children allocated to the Ventriloquist Puppet group (Active Comparator): Children allocated to the Ventriloquist Puppet group were introduced to a Ventriloquist Puppet inside the clinic and were allowed to play , talk and interact with the puppet for five to 10 min
  Interventions: Behavioral: Ventriloquist Puppet Interaction

INTERVENTIONS:
Behavioral: Ventriloquist Puppet Interaction — children allocated to the Ventriloquist Puppet group were introduced to a Ventriloquist Puppet inside the clinic and were allowed to play, talk, and interact with the puppet for 5-10 minutes.
  Arms: puppet therapy group: Children allocated to the Ventriloquist Puppet group

SUMMARY:
thhe goal of this clinical trial is to assess the effect of ventriloquist puppets to reduce the strees accompined by the dental visit in cgilren . The main questions it aims to answer are:

* Does the ventriloquist puppet can reduce the stress accompanied by the dental visit for the children ?
* What medical problems do participants have when taking drug ABC? Researchers will compare ventriloquist puppet to a control group (conventional behavior management techniques ) to see if ventriloquist puppet can lower the anxiety or not.

ELIGIBILITY:
Inclusion Criteria :

* healthy children with no systemic diseases.
* children require dental intervention

Exclusion Criteria:

* children with bad dental experience
* children require invasive surgical intervention

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Dental anxiety | From immediately before to immediately after the dental procedure
  Change in Anxiety Score using MCDAS scale
Heart rate | From immediately before to immediately after the dental procedure
  change in heart rate during the visit to investigate the anxiety effect using pulse oximeter

IPD SHARING:
Plan to Share IPD: No